CLINICAL TRIAL: NCT00003456
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Glioblastoma Multiforme
Brief Title: Antineoplaston Therapy in Treating Patients With Newly-diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066488; BRI-BT-07 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: adult glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a newly diagnosed Glioblastoma Multiforme will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for Glioblastoma Multiforme provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults (≥ 18 years of age) with newly diagnosed Glioblastoma Multiforme.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which adults (≥ 18 years of age) with newly diagnosed Glioblastoma Multiforme receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults (≥ 18 years of age) with newly diagnosed Glioblastoma Multiforme, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults (≥ 18 years of age) with newly diagnosed Glioblastoma Multiforme.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed Glioblastoma Multiforme
* Subtotal resection or biopsy only of tumor
* Measurable tumor by MRI scan performed within two weeks prior to study entry
* Tumor must be at least 5 mm
* No brain stem tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 4 months

Hematopoietic:

* WBC at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* No hepatic failure
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that would contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No concurrent immunomodulatory agents

Chemotherapy:

* No prior chemotherapy
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from any prior surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1995-03-14 (Actual); Primary Completion 2004-12-07 (Actual); Study Completion 2004-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty patients were recruited between March 1995 and June 2004. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Adults with a newly diagnosed Glioblastoma Multiforme will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 40
Completed | 32
Not Completed | 8
Not completed — Not evaluable | 8

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 52.4 [26.3 to 76.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 32
Participants
  Complete Response | 2
  Partial Response | 1
  Stable Disease | 2
  Progressive Disease | 27

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Percentage of participants
  6 months overall survival | 27.5
  12 months overall survival | 12.5
  24 months overall survival | 7.5
  36 months overall survival | 5.0
  48 months overall survival | 2.5
  60 months overall survival | 2.5

ADVERSE EVENTS:
Time Frame: 9 years, 6 months
Description: Forty patients were recruited between March 1995 and December 2004. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Central venous catheter: Infection (General disorders) | 1 — The Central venous catheter: Infection was not related to Antineoplaston therapy.
The Central venous catheter: Thrombosis/embolism. (General disorders) | 1 — The Central venous catheter: Thrombosis/embolism was not related to Antineoplaston therapy.
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 — The Fatigue (asthenia, lethargy, malaise) was not related to Antineoplaston therapy.
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 — The Injection site reaction/extravasation changes was/were not related to Antineoplaston therapy.
Vomiting (Gastrointestinal disorders) | 1 — The Vomiting was not related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 1 — The Hemorrhage, CNS was not related to Antineoplaston Therapy.
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 1 — The Infection (documented clinically): Bladder (urinary) was not related to Antineoplaston Therapy.
Lung (pneumonia) (Infections and infestations) | 1 — The Lung (pneumonia) was not related to Antineoplaston Therapy
Hypernatremia (Investigations) | 2 — One of the Hypernatremias was related to Antineoplaston Therapy. One of the Hypernatremias was not related to Antineoplaston Therapy.
Seizure (Nervous system disorders) | 2 — The Seizures were not related to Antineoplaston Therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 7 — The Somnolences/depressed levels of consciousness were not related to Antineoplaston Therapy.
Syncope (fainting) (Nervous system disorders) | 1 — The Syncope (fainting) was not related to Antineoplaston Therapy.
Pain: Head/headache (Nervous system disorders) | 3 — The Pain: Head/headaches were not related to Antineoplaston Therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 — The Dyspneas (shortnesses of breath) were not related to Antineoplaston Therapy.
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 — The Pleural effusion (non-malignant) was not related to Antineoplaston Therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 2 — The Thromboses/thrombi/embolisms were not related to Antineoplaston Therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 10
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 7
Hypertension (Cardiac disorders) | 2
Central Venous Catheter: Infection (General disorders) | 4
Central Venous Catheter: Non-functional (General disorders) | 7
Central Venous Catheter: Other (General disorders) | 4
Central Venous Catheter: Pain (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 28
Fever (General disorders) | 6
Edema/Fluid retention (General disorders) | 15
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 11
Hemorrhage, GU (Renal and urinary disorders) | 2
Infection (documented clinically): Bladder (urinary) (Renal and urinary disorders) | 4
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Mucosa (Infections and infestations) | 3
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 5
Infection: Upper airway (Infections and infestations) | 2
Hyperbilirubinemia (Investigations) | 2
Hyperglycemia (Investigations) | 12
Hypernatremia (Investigations) | 17
Hypocalcemia (Investigations) | 3
Hypoglycemia (Investigations) | 8
Hypokalemia (Investigations) | 25
Proteinuria (Investigations) | 2
SGOT (Investigations) | 7
SGPT (Investigations) | 9
Ataxia (incoordination) (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 10
Neuropathy: motor (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 7
Somnolence/depressed level of consciousness (Nervous system disorders) | 21
Speech impairment (Nervous system disorders) | 8
Pain: Head/headache (Nervous system disorders) | 16
Pain: Joint (Musculoskeletal and connective tissue disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Thrombosis/thrombus/embolism 1 2 3 (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No